CLINICAL TRIAL: NCT01853085
Title: A Study of Patients With Primary Open Angle Glaucoma or Ocular Hypertension Switched to Lumigan® UD Monotherapy for Medical Reasons
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/038
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with POAG or OHT: Patients with primary open angle glaucoma (POAG) or ocular hypertension (OHT) treated with Lumigan® UD (bimatoprost ophthalmic solution) administered in accordance with physician standard practice for up to 12 weeks.
  Interventions: Drug: Bimatoprost Ophthalmic Solution

INTERVENTIONS:
Drug: Bimatoprost Ophthalmic Solution — Patients with primary open angle glaucoma (POAG) or ocular hypertension (OHT) treated with Lumigan® UD (bimatoprost ophthalmic solution) administered in accordance with physician standard practice for up to 12 weeks.
  Other Names: Lumigan® UD

SUMMARY:
The study will evaluate patients diagnosed with primary open angle glaucoma or ocular hypertension who are switched to Lumigan® UD monotherapy for medical reasons in accordance with physician standard clinical practice. All treatment decisions lie with the physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma or ocular hypertension
* Previously prescribed intraocular pressure (IOP)-lowering medication with insufficient IOP control and is now being switched to Lumigan® UD for medical reasons

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary open-angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 1830 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Wiesloch, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Pillunat LE, Eschstruth P, Hasemeyer S, Thelen U, Foja C, Leaback R, Pfennigsdorf S. Preservative-free bimatoprost 0.03% in patients with primary open-angle glaucoma or ocular hypertension in clinical practice. Clin Ophthalmol. 2016 Sep 12;10:1759-65. doi: 10.2147/OPTH.S103084. eCollection 2016. PMID 27672307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With POAG or OHT
Started | 1830
Completed | 1595
Not Completed | 235

BASELINE CHARACTERISTICS:
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1830
Age, Customized [Number; unit: Participants]
  <18 years | 1
  18-30 years | 9
  31-40 years | 28
  41-50 years | 130
  51-60 years | 328
  61-70 years | 509
  71-80 years | 601
  81-90 years | 158
  ≥ 91 years | 16
  Missing Data | 50
Sex/Gender, Customized [Number; unit: Participants]
  Female | 1098
  Male | 723
  Missing Data | 9

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) in the Study Eye at Baseline
Description: IOP is a measurement of the fluid pressure inside the study eye.
Time Frame: Baseline
Population: All patients with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1672
Millimeters of Mercury (mmHg) | 21.15 (3.43)

2. Secondary Outcome: Physician Assessment of IOP-Lowering Effect in the Study Eye on a 3-Point Scale
Description: IOP is a measurement of the fluid pressure inside the eye. Physicians evaluate IOP change from baseline in the study eye as better than expected, as expected, and worse than expected. The numbers of patients in each category are presented.
Time Frame: Baseline, 12 Weeks
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1716
Patients
  Better than Expected | 649
  As Expected | 916
  Worse than Expected | 151

3. Secondary Outcome: Patient Assessment of Tolerability on a 4-Point Scale
Description: Patient assessment of tolerability is assessed using a 4-point scale (very good, good, moderate, and poor). The numbers of patients in each category are presented.
Time Frame: 12 Weeks
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1730
Patients
  Very Good | 913
  Good | 670
  Moderate | 73
  Poor | 74

4. Secondary Outcome: Physician Assessment of Tolerability on a 4-Point Scale
Description: Physician assessment of tolerability is assessed using a 4-point scale (very good, good, moderate, and poor). The numbers of patients in each category are presented.
Time Frame: 12 Weeks
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1746
Patients
  Very Good | 982
  Good | 648
  Moderate | 78
  Poor | 38

5. Secondary Outcome: Number of Patients Who Discontinue Treatment With Lumigan® UD Prior to 12 Weeks of Treatment
Description: Patient discontinuation of treatment with Lumigan® UD prior to 12 weeks of treatment is assessed as Yes or No.
Time Frame: 12 Weeks
Population: All enrolled patients
Measure: Number; unit: Patients
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1830
Patients | 139

6. Secondary Outcome: Number of Patients Who Continue Treatment
Description: Patient continuation of treatment with Lumigan® UD after the end of study participation is assessed as Yes or No.
Time Frame: 12 Weeks
Population: All enrolled patients
Measure: Number; unit: Patients
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1830
Patients | 1501

7. Secondary Outcome: Physician Assessment of Patient Compliance Compared to Previous Treatment on a 3-Point Scale
Description: Physician assessment of patient compliance compared to previous therapy is assessed on a 3-point scale (better, equal, and worse). The numbers of patients in each category are presented.
Time Frame: 12 Weeks
Population: All patients with data for this outcome measure
Measure: Number; unit: Patients
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1675
Patients
  Better | 848
  Equal | 777
  Worse | 50

8. Primary Outcome: IOP in the Study Eye at Week 12
Description: IOP is a measurement of the fluid pressure inside the study eye.
Time Frame: Week 12
Population: All patients with data for this outcome measure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 1672
mmHg | 16.38 (2.93)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for 12 weeks.
Arm/Group | Patients With POAG or OHT
Serious Adverse Events (participants affected / at risk) | 2/1830
Other Adverse Events (participants affected / at risk) | 0/1830
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With POAG or OHT (N=1830)
Cataract Operation (Eye disorders) | 1
Death (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.